CLINICAL TRIAL: NCT05268146
Title: Characterization, Creativity, Leadership, and Search for Solutions to Improve the Lifestyles of Earlier Elderly People in Urban Areas
Brief Title: Earlier Elderly People in Urban Areas
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Rosa Sola, Full Professor, Dr., University Rovira i Virgili
Other Study IDs: Earlier-Elderly Urban People
Record Dates: First submitted 2022-02-11; First posted 2022-03-07 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenia; Eldery People; Lifestyle, Healthy; Nutrition; Sleep; Physical Activity; Participatory Research
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lifestyles — Co-creation process and participatory research; lifestyles

SUMMARY:
Social innovation in aging needs to bring new ideas and services to meet new social and welfare needs identified in recent years. In our environment, people ≥60 years old accounted for 20% -24% of the population in 2015, and it is expected to increase to ≥30% by 2050.

The objectives of this project are: To characterize the elderly (60 to 74 years) who live independently in urban areas of the province of Tarragona, to actively involve them, through a process of participatory research to generate solutions.

To achieve this goal, it is proposed to make a diagnosis of their health status (lifestyles, risk of malnutrition, and sarcopenia), and conduct focus groups including young seniors from urban areas, and stakeholders, to determine their needs, interests, and barriers for pursuing healthy lifestyles. Based on the information obtained in the diagnosis and focus groups, there will be processes for co-creating solutions based on proposed activities or changes in their immediate environment.

DETAILED DESCRIPTION:
Social innovation in aging needs to bring new ideas and services to meet new social and welfare needs identified in recent years. In our environment, people ≥60 years old accounted for 20% -24% of the population in 2015, and it is expected to increase to ≥30% by 2050. For the first time in history, most people can aspire to live well beyond the age of 60. On the other hand, the Covid-19 pandemic has severely affected people ≥60 years of age and may make the welfare and health problems of this population more evident, such as unhealthy lifestyles, the risk of malnutrition, and sarcopenia (defined as loss of muscle mass, strength, and function), which leads to significant dependency and quality of life problems. In addition, older people living in urban areas have been severely affected by confinement, and new needs are being generated. To better understand the needs, an innovative element of this project is to involve the elderly-young people (60-74 years) from urban areas in the generation of solutions, which will make these solutions especially adapted to their needs. Therefore increase the adherence to the solutions created, and also the long-term sustainability of the solutions.

The objectives of this project are: To characterize the elderly (60 to 74 years) who live independently in urban areas of the province of Tarragona, to actively involve them, through a process of participatory research to generate solutions.

To achieve this goal, it is proposed to make a diagnosis of their health status (lifestyles, risk of malnutrition, and sarcopenia), and conduct focus groups including young seniors from urban areas, and stakeholders, to determine their needs, interests, and barriers for pursuing healthy lifestyles. Based on the information obtained in the diagnosis and focus groups, there will be processes for co-creating solutions based on proposed activities or changes in their immediate environment. During the co-creation process, the elderly and the 4-helix stakeholders (government, industry, university, and civil society) will be involved.

ELIGIBILITY:
Inclusion Criteria:

* People ≥60 years and ≤75 years,
* That they have informed consent,
* Living at home (living independently), Community-dwelling early-elderly
* That they can continue the study,
* They live in the province of Tarragona

Exclusion Criteria:

* Failure to comply with the inclusion criteria will be considered an exclusion criterion.

Ages: 60 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Earlier elderly people living in urban areas. The target population will be recruited from different places in the community, town halls, civic centers, senior citizens' associations, etc.
Sampling Method: Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Risk of sarcopenia (muscle strength) | 1 day
  Reduction of muscle strength: <27kg in men and <16kg in women measured by a dynamometer
Diagnosis of sarcopenia (muscle strength) | 1 day
  Reduction of muscle strength (<27kg in men and <16kg in women measured by a dynamometer)
Diagnosis of sarcopenia (muscle mass) | 1 day
  Reduction of muscle mass (<20kg in men and <15kg in women measured by bioimpedance)
Diagnosis of severe sarcopenia (muscle strength) | 1 day
  Reduction of muscle strength (<27kg in men and <16kg in women measured by a dynamometer) and
Diagnosis of severe sarcopenia (muscle mass) | 1 day
  Reduction of muscle mass (<20kg in men and <15kg in women measured by bioimpedance)
Diagnosis of severe sarcopenia (muscle function) | 1 day
  Reduction of muscle function (≤0.8 m / s)

SECONDARY OUTCOMES:
Nutrition | 1 day
  Food frequency questionnaire
  (not scale)
Physical activity | 1 day
  International physical activity questionnaire for elderly Low category: non-physical activity or it is not enough to achieve moderate or high category Moderate category: 3 or more days / weeks (vigorous physical activity, at least 25 minutes/day), or 5 or more (moderate physical activity, at least 30 minutes/day), or 5 or more days / weeks of a combination of walking, or moderate-vigorous physical activity (at least 600 METS).
  High category: 7 or more days / week of a combination of walking, or moderate-vigorous physical activity (at least 3000 METS).
Sleep behaviour | 1 day
  Pittsburg questionnaire
  Pittsburg questionnaire The questionnaire contains a total of 19 questions, grouped into 10 questions. The 19 questions are combined to form seven areas with their corresponding score, each of which shows a range between 0 and 3 points. In all cases, a score of "0" indicates ease, while a score of 3 indicates severe difficulty, within their respective area. The score of the seven areas is finally added to give an overall score, which ranges from 0 to 21 points. "0" indicates ease of sleeping and "21" severe difficulty in all areas.
Risk of malnutrition | 1 day
  Mini Nutritional Assessment 12-14 points: normal nutritional status 8-11 points: risk of malnutrition 0-7 points: malnutrition
Weight | 1 day
  Weight using a balance (kg)
height | 1 day
  Height using a tallimeter (m)
BMI | 1 day
  Using weight (kg) / height (m)2

OTHER OUTCOMES:
Age | 1 day
  Age in years
Gender | 1 day
  Female or male

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Sola, Dr, Principal Investigator — University Rovira i Virgili
Locations (2):
- Spain (2):
  - Institut d'Investigació Sanitaria Pere i Virgili, Reus, Tarragona
  - University Rovira i Virgili, Reus, Tarragona

IPD SHARING:
Plan to Share IPD: No